CLINICAL TRIAL: NCT00741923
Title: Beans and Potatoes in the Regulation of Food Intake and Risk Factors for Chronic Diseases. Effect of Consuming Beans for One Month on Blood Lipids, Satiety, Intake Regulation and Body Weight
Brief Title: Effect of Consuming Beans for One Month on Blood Lipids, Satiety, Intake Regulation and Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ontario Ministry of Agriculture, Food and Rural Affairs (Other Government)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OMAF-HEINZbeans; BOW-2008
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Overweight; Obesity; Metabolic Syndrome; Diabetes; Hypertension
Keywords: beans; pulses; satiety; appetite; obesity; overweight; diabetes; metabolic syndrome; hypertension; blood glucose; insulin; cholesterol; HDL; LDL; leptin; GLP-1; adiponectin; Peptide YY; diet
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Diabetes Mellitus; Hypertension; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bean group (Experimental): A group consuming 5 cups/week of navy beans for a month
  Interventions: Other: navy beans added to regular diet

INTERVENTIONS:
Other: navy beans added to regular diet — 5 cups per week of commercially available white beans for 4-weeks
  Other Names: Heinz beans

SUMMARY:
This project investigates the effect of regular consumption of commercially available processed white beans (5 cups per week) on food intake, body weight, blood pressure, satiety hormones and glycemic response over a 4-week period. We have chosen to provide participants with canned white beans, the most accessible and frequently consumed bean in North America. They are inexpensive, a good source of high quality nutrients and ready to eat. Based upon published literature and short-term studies conducted in our laboratory, we hypothesize that regular consumption of commercially available canned beans will increase satiety and improve the control of food intake, body weight, blood glucose and blood lipids.

DETAILED DESCRIPTION:
The metabolic syndrome is a clustering of chronic disease risk factors, including abdominal obesity, dyslipidemia, elevated blood pressure and elevated fasting blood glucose.

A main treatment for metabolic syndrome is lifestyle modification (alterations in diet and/or physical activity patterns) resulting in weight loss.

Beans are easily incorporated into the diet and may lead to the attainment and maintenance of healthy a body weight and improved metabolic control.

Canned baked navy beans (with tomato sauce) have a low glycemic response following consumption, however, whether this effect has long-term benefits on glycemic control requires further investigation.

OBJECTIVE

To determine the effect of consuming 5 cups per week of commercially available canned navy beans over 4 weeks on risk factors associated with the metabolic syndrome.

Subjects

Inclusion criteria: Men and women (n=16) between 35 and 55 years of age with a body mass index (BMI) of 27 to 40 kg/m2.

Exclusion criteria: smoking or any major surgery/medical condition within the last 6 months, use of medications that could interfere with the study outcomes, gastrointestinal, liver or kidney disease and women who were pregnant/lactating

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-40 kg/m2

Exclusion Criteria:

* smokers and individuals who have prescribed medications over the past 6 months that could interfere with the study outcomes (i.e. statins, metformin). Breakfast skippers, those on a restricted energy diet or pregnant/lactating women

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
body weight, waist circumference, blood glucose, satiety hormones, and blood lipids, inflammation factor, and glycated haemoglobin | at the beginning and at the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, Ph.D., Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, University of Toronto, Toronto, Ontario, Canada